CLINICAL TRIAL: NCT04615403
Title: Prospective, Non-Randomized, Open-Label, Multi-Center, Single Arm Study of Exchange of Travoprost Intraocular Implant
Brief Title: Study of Exchange of Travoprost Intraocular Implant
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Glaukos Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IDOS-106-EXCH
Record Dates: First submitted 2020-10-29; First posted 2020-11-04 (Actual); Results first posted 2023-09-26 (Actual); Last update posted 2023-09-26 (Actual); Status verified 2023-09

CONDITIONS: Open Angle Glaucoma
MeSH Terms: conditions — Glaucoma, Open-Angle | interventions — Travoprost

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Implantation and Exchange (Experimental): Subjects will undergo implantation and exchange of a Travoprost Intraocular Implant through a small temporal clear corneal incision.
  Interventions: Drug: Travoprost

INTERVENTIONS:
Drug: Travoprost — Implantation and exchange of a Travoprost Intraocular Implant through a clear corneal incision

SUMMARY:
The study objective is to evaluate the safety of the operative and surgical exchange procedure of Travoprost Intraocular Implant in subjects with open-angle glaucoma or ocular hypertension.

DETAILED DESCRIPTION:
This prospective, non-randomized, open-label, multi-center, single arm, clinical trial intends to implant approximately 45 male and female subjects over 18 years old who have been diagnosed with open-angle glaucoma (OAG) or ocular hypertension (OHT). All subjects are required to meet eligibility criteria at Visit 1 (Screening). The purpose of this study is to evaluate the safety of the implantation and exchange of a Travoprost Intraocular Implant in subjects with open-angle glaucoma or ocular hypertension. Postoperatively, there are 6 follow-up visits over a 12 month period.

ELIGIBILITY:
Inclusion Criteria:

* Able and willing to attend scheduled follow-up exams for the duration of the study
* Able and willing to provide written informed consent on the IRB (institutional review board)/IEC (institutional ethics committee)-approved Informed Consent form
* Best spectacle corrected visual acuity of 20/80 or better in each eye.
* Previously qualified for GC-009 clinical trial using the Travoprost Intraocular Implant with the travoprost intraocular implant (G2TR) that is present in the study eye.

Exclusion Criteria:

* Glaucoma status as follows:

  * Traumatic, uveitic, neovascular, or angle-closure glaucoma; or glaucoma associated with vascular disorders
* Corneal status as follows:

  * Any active inflammation or edema
* Any pathology for which, in the investigator's judgement, the following would be either at risk or contraindicated:
* Implantation of Travoprost Intraocular Implant
* Compliance to elements of the study protocol (e.g., ophthalmic examinations, follow-up visits)
* Fellow eye status as follows:

  * Fellow eye actively enrolled in this trial or any other clinical trial
* Subject status as follows:

  * Pregnant or planning to become pregnant during the course of the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2020-11-19 (Actual); Primary Completion 2022-02-28 (Actual); Study Completion 2022-02-28 (Actual)

CONTACTS AND LOCATIONS:
Locations (14):
- United States (13):
  - Inland Eye Specialists, Hemet, California
  - North Bath Eye Associates, Inc., Petaluma, California
  - Eye Center of northern Colorado, PC, Fort Collins, Colorado
  - The Eye Associates of Manatee, Manatee, Florida
  - Ocala Eye, Ocala, Florida
  - Center for Sight, Sarasota, Florida
  - Jones Eye Clinic, Sioux City, Iowa
  - D'Ambrosio Eye Care, Lancaster, Massachusetts
  - Northern New Jersey Eye Institute, South Orange, New Jersey
  - Oklahoma Eye Surgeons, Oklahoma City, Oklahoma
  - Vance Thompson Vision, Sioux Falls, South Dakota
  - Texan Eye, Austin, Texas
  - Lehmann Eye Center, Nacogdoches, Texas
- Asian Eye Institute, Makati City, Philippines

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Implantation and Exchange
Started | 33
Completed | 32
Not Completed | 1
Not completed — Death | 1

BASELINE CHARACTERISTICS:
Population: safety population (all participants who underwent the exchange procedure)
Arm/Group | Implantation and Exchange
Number analyzed (Participants) | 33
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 15
  >=65 years | 18
Age, Continuous [Mean (Standard Deviation); unit: years] | 65.2 (11.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17
  Male | 16
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2
  Not Hispanic or Latino | 31
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 2
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 28
  More than one race | 0
  Unknown or Not Reported | 1
Duration since initial implant administration [Mean (Standard Deviation); unit: days] — time (days) since the administration of the previous travoprost intraocular implant
  days | 1540.8 (123.7)

OUTCOME MEASURES:

1. Primary Outcome: Ocular Safety
Description: Number of subjects with Adverse Events including intra-operative and post-operative events (TEAE's) in the study eye
Time Frame: 12 Months
Population: Safety population (all subjects who underwent the exchange procedure)
Measure: Number; unit: subjects
Arm/Group | Implantation and Exchange
Number analyzed (Participants) | 33
subjects | 13

ADVERSE EVENTS:
Time Frame: 12 months
Arm/Group | Implantation and Exchange
All-Cause Mortality (participants affected / at risk) | 1/33
Serious Adverse Events (participants affected / at risk) | 2/33
Other Adverse Events (participants affected / at risk) | 16/33
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Implantation and Exchange (N=33)
Death (General disorders) | 1 (1) — Death of unknown cause
Retinal vein occlusion (Eye disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Implantation and Exchange (N=33)
Eye irritation (Eye disorders) | 2 (2)
Corneal pigmentation (Eye disorders) | 1 (1)
Diabetic retinopathy (Eye disorders) | 1 (2) — 1 event in study eye, 1 event in fellow eye
Iridodialysis (Eye disorders) | 1 (1)
Photophobia (Eye disorders) | 1 (1)
Posterior capsule opacification (Eye disorders) | 1 (2) — 1 event in study eye, 1 event in fellow eye
Retinal hemorrhage (Eye disorders) | 1 (1)
Hordeolum (Eye disorders) | 1 (1)
Conjunctivitis viral (Eye disorders) | 1 (1) — non-study eye AE
Corneal abrasion (Eye disorders) | 1 (1)
Corona virus infection (Infections and infestations) | 2 (2)
Ear infection (Infections and infestations) | 1 (1)
Gout (Metabolism and nutrition disorders) | 1 (1)
Atonic seizures (Nervous system disorders) | 1 (1)
Cerebral arteriosclerosis (Nervous system disorders) | 1 (1)
Trigeminal neuralgia (Nervous system disorders) | 1 (1)
Visual field defect (Nervous system disorders) | 3 (3)
Intraocular pressure increased (Investigations) | 2 (2)

LIMITATIONS AND CAVEATS:
This was a single arm, open label study in a small number of subjects to assess safety of administration of a second implant and removal of the previous implant.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor reserves the right of prior review of any publication or presentation of data from this study.

DOCUMENTS (2):
  • Study Protocol (2020-08-24): https://cdn.clinicaltrials.gov/large-docs/03/NCT04615403/Prot_000.pdf
  • Statistical Analysis Plan (2022-03-02): https://cdn.clinicaltrials.gov/large-docs/03/NCT04615403/SAP_001.pdf